CLINICAL TRIAL: NCT00656643
Title: A Phase 2, Randomized, Double-Masked, Placebo-Controlled, Dose-Ranging Clinical Study to Assess the Safety and Efficacy of Subconjunctival Injections of Sirolimus in Patients With Diabetic Macular Edema Secondary to Diabetic Retinopathy
Brief Title: Dose Ranging Study of an Ocular Sirolimus (Rapamycin) Formulation in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: MacuSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR-002
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2010-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Sirolimus
- 2 (Experimental)
  Interventions: Drug: Sirolimus
- 3 (Experimental)
  Interventions: Drug: Sirolimus
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Two subconjunctival injections of 440 micrograms sirolimus each.
  Other Names: MS-R001, rapamycin
  Arms: 2
Drug: Placebo — Two subconjunctival injections of placebo.
  Other Names: Vehicle
  Arms: 4
Drug: Sirolimus — Two subconjunctival injections of 220 micrograms sirolimus each.
  Other Names: MS-R003, rapamycin
  Arms: 1
Drug: Sirolimus — Two subconjunctival injections of 880 micrograms sirolimus each.
  Other Names: MS-R002, rapamycin
  Arms: 3

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an ocular sirolimus (rapamycin) formulation at various doses in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria include but are not limited to:

* Diagnosed with diabetes mellitus
* Macular edema secondary to diabetic retinopathy
* Visual acuity of 20/40 to 20/200 in study eye

Exclusion Criteria include but are not limited to:

* Any other ocular disease that could compromise vision in the study eye
* Any of the following treatments to the study eye within 90 days prior to study start: intravitreal injections; posterior subtenons steroids; focal/grid macular photocoagulation; intraocular surgery
* Capsulotomy of the study eye within 30 days prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity by ETDRS | 180 days

SECONDARY OUTCOMES:
Foveal central subfield thickness as determined by OCT | 180 days
Safety across dose groups versus placebo | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, MD, Study Director — MacuSight, Inc.
Locations (1):
- Retinal Consultants of Arizona, Phoenix, Arizona, United States